CLINICAL TRIAL: NCT00867217
Title: A Randomized Trial to Evaluate the Benefit of High Dose Vitamin D3 on Aromatase Inhibitor Letrozole-Associated Musculoskeletal Symptoms and Fatigue (The VITAL Trial).
Brief Title: Vitamin D3 for Aromatase Inhibitor Induced Arthralgias
Acronym: VITAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Qamar Khan (Other)
Collaborators: Novartis Pharmaceuticals (Industry); BTR Group (Industry)
Responsible Party: Sponsor-Investigator, Qamar Khan, Associate Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 11548
Record Dates: First submitted 2009-03-20; First posted 2009-03-23 (Estimated); Results first posted 2018-02-09 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Vitamin D; Cholecalciferol; Letrozole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Dose Vitamin D (Experimental): High Dose Vitamin D3 capsule (3 x 10,000 IU capsules weekly). All subjects also received standard dose vitamin D3 (600 IU daily) and letrozole (2.5 mg daily).
  Interventions: Dietary Supplement: High Dose Vitamin D; Dietary Supplement: Standard Dose Vitamin D3; Drug: Letrozole 2.5mg
- Placebo (Placebo Comparator): Placebo matched for High Dose Vitamin D3 capsules. All subjects also received standard dose vitamin D3 (600 IU daily) and letrozole (2.5 mg daily).
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Standard Dose Vitamin D3; Drug: Letrozole 2.5mg

INTERVENTIONS:
Dietary Supplement: High Dose Vitamin D — High Dose Vitamin D3 (3 capsules of 10,000 IU) weekly for 24 weeks.
  Arms: High Dose Vitamin D
Dietary Supplement: Placebo — Placebo comparator
  Arms: Placebo
Dietary Supplement: Standard Dose Vitamin D3 — Standard Dose Vitamin D3 (600 IU of vitamin D3 daily)
Drug: Letrozole 2.5mg — All subjects received letrozole as standard of care.

SUMMARY:
The primary purpose is to determine if high dose vitamin D3 reduces the incidence of musculoskeletal symptoms associated with the aromatase inhibitor letrozole in women with early stage breast cancer and low serum vitamin D levels.

DETAILED DESCRIPTION:
The primary hypothesis is that high dose vitamin D3 plus standard dose vitamin D3 prevents the worsening of musculoskeletal symptoms when compared to a standard dose vitamin D3 treatment. This protocol will examine the relationship between vitamin D levels (25-hydroxyvitamin D) and various quality of life measures in women being treated with letrozole as standard care for early stage breast cancer. All subjects received letrozole and a standard dose of vitamin D3 (600 IU daily). Randomization was between high dose vitamin D3 (30,000 IU once per week) vs. a blinded, matched placebo,

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women newly diagnosed with early stage breast cancer, who would be treated with an aromatase inhibitor
* Serum 25OHD levels < 40 ng/ml

Exclusion Criteria:

* Severe or debilitating musculoskeletal pain
* Known metastatic disease
* History of renal stones
* History of hypercalcemia or hyperthyroidism
* Currently receiving adjuvant or neoadjuvant chemotherapy
* Currently receiving other investigational agents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2009-03; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Qamar J Khan, MD, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - University of Kansas Medical Center, Westwood, Kansas
  - Cancer Centers of Kansas, P.A., Wichita, Kansas

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo (3 capsules of matching placebo given weekly) along with standard of care medication (Standard Dose Vitamin D3, 600 IU of vitamin D3 daily; letrozole, 2.5 mg daily) for 24 weeks.
- Vitamin D: High Dose Vitamin D3 (3 capsules of 10,000 IU given weekly) along with standard of care medication (Standard Dose Vitamin D3, 600 IU of vitamin D3 daily; letrozole, 2.5 mg daily) for 24 weeks.
Period: Overall Study
Arm/Group | Placebo | Vitamin D
Started | 80 | 80
Completed | 77 | 70
Not Completed | 3 | 10

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo (3 capsules of matching placebo weekly) along with standard of care medication (Standard Dose Vitamin D3, 600 IU of vitamin D3 daily; letrozole, 2.5 mg daily) for 24 weeks.
- Vitamin D: High Dose Vitamin D3 (3 capsules of 10,000 IU weekly) along with standard of care medication (Standard Dose Vitamin D3, 600 IU of vitamin D3 daily; letrozole, 2.5 mg daily) for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Vitamin D | Total
Number analyzed (Participants) | 80 | 80 | 160
Age, Customized [Median (Full Range); unit: years] | 62 [34 to 87] | 60.5 [42 to 85] | 62 [34 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 80 | 160
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 75 | 77 | 152
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 80 | 80 | 160

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Worsening of Musculoskeletal Symptoms (MS)
Description: Worsening of Musculoskeletal Symptoms (MS) is defined as any one of the following three events: (a) an increase by at least 0.25 in the Health Assessment Questionnaire II (HAQ II, a measure of disability from joint pain) score, (b) an increase in patient reported severity of joint and/or muscle pain, or (c) discontinuation from trial prior to 24 weeks specifically because of problems with musculoskeletal symptoms.
Time Frame: Change from Baseline to 24 Weeks
Population: Subjects available for analysis included those that had completed the entire study; plus three subjects that had dropped out early specifically because of side effects related to musculoskeletal symptoms (one of the endpoints).
Measure: Number; unit: participants
Groups:
- Placebo: Placebo (3 capsules of matching placebo) along with standard of care medication (Standard Dose Vitamin D3; 600 IU of vitamin D3 daily) given weekly for 24 weeks
- Vitamin D: High Dose Vitamin D3 (3 capsules of 10,000 IU) capsules along with standard of care medication standard of care medication (Standard Dose Vitamin D3; 600 IU of vitamin D3 daily) given weekly for 24 weeks
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 77 | 70
participants
  HAQ II increase by 0.25 | 23 | 18
  Subjective Pain increase | 24 | 18
  Discontinuation due to AEs | 3 | 0
  Any of the three measures | 39 | 26

ADVERSE EVENTS:
Time Frame: 1 year, 9 months
Description: Adverse events were collected either at routine clinical visits or by patient report during periodic phone calls.
Groups:
- Vitamin D: High Dose Vitamin D3 (3 capsules of 10,000 IU) capsules along with standard of care medication standard of care medication (Standard Dose Vitamin D3; 600 IU of vitamin D3 daily) given weekly
Arm/Group | Placebo | Vitamin D
Serious Adverse Events (participants affected / at risk) | 3/80 | 3/80
Other Adverse Events (participants affected / at risk) | 67/80 | 37/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=80) | Vitamin D (N=80)
Cardiac Changes (Cardiac disorders) | 0 | 1
CNS Ischemia (Nervous system disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Hemolysis (Blood and lymphatic system disorders) | 1 | 0
Supraventricular arryhthmia (Cardiac disorders) | 0 | 1
Wound Complications (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=80) | Vitamin D (N=80)
Arthralgia (Nervous system disorders) | 4 | 7
Fatigue (Nervous system disorders) | 9 | 6
Hot Flashes (General disorders) | 12 | 3
Joint Function (Musculoskeletal and connective tissue disorders) | 9 | 10
Joint Pain (Musculoskeletal and connective tissue disorders) | 16 | 6
Nausea (Gastrointestinal disorders) | 3 | 5
Pain - Back (Nervous system disorders) | 4 | 3
Pain - Hip (Nervous system disorders) | 5 | 1
Pain - Shoulder (Nervous system disorders) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes